CLINICAL TRIAL: NCT03229902
Title: A Non-Concurrent, Multiple-Baseline, Across-Subjects Trial of Mantra Meditation in Subjects That Have Chronically Impaired Attention After Stroke
Brief Title: Mantra Meditation in Subjects That Have Chronically Impaired Attention After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cheryl Carrico (Other)
Responsible Party: Sponsor-Investigator, Cheryl Carrico, principal investigator, University of Kentucky
Organization: University of Kentucky (Other)
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 170013F6A
Record Dates: First submitted 2017-07-20; First posted 2017-07-26 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Stroke Sequelae
Keywords: stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: single-case research design involving a series of AB designs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mantra meditation (Experimental): Each session of mantra meditation lasts for 30 minutes. The participants in each session comprise 1 subject and the PI. In each session, the subject and the PI co-participate in repetitive intonation of a pre-specified mantra. Intervention is comprised of 9 sessions, each of which occurs on a separate weekday at approximately equal intervals over a total intervention period of 3 weeks.
  Interventions: Behavioral: mantra meditation

INTERVENTIONS:
Behavioral: mantra meditation — see study description

SUMMARY:
There is an evidence gap on whether meditation may improve behaviorally measured attention after stroke, but preliminary research is promising. This study is the first-ever investigation of whether mantra meditation may improve chronic, severe impairment in attention after stroke.

DETAILED DESCRIPTION:
The study is non-concurrent, multiple-baseline, across-subjects, single-case research design (SCRD). The central hypothesis is that mantra meditation (independent variable) will be associated with improvement on 1 or more tests of behaviorally measured sustained attention (dependent variable). The mantra in this study is the syllable "um" and is not assigned any spiritual, religious, or affective meaning. The mantra is repeated aloud together by the subject and the PI for a duration of 30 minutes in each session. This procedure constitutes meditation for the purposes of this study. There are 9 session of meditation (3 times per week for 3 weeks). Attention is measured in each of these sessions as well as in 3 separate testing sessions that precede the intervention period.

ELIGIBILITY:
Inclusion Criteria.

1. Adults between the ages of 18 and 70
2. Chronic, non-lacunar, right-hemisphere stroke (i.e., sustained at >12 months prior to date of clinical screen)
3. Severely impaired attention defined as 5 or more errors of commission on the SARTfixed
4. Intact consent capacity with no evidence of dementia, defined as a score of 100% correct answer rate on University of California, San Diego Brief Assessment of Capacity to Consent (UBACC).
5. Right-handed dominance as well as sufficient movement and vision function for testing (use of computer mouse, keyboard, and monitor)
6. English language fluency and reading comprehension at least at 6th grade level

Exclusion Criteria.

1. Depression defined as a score of >10 on Beck Depression Inventory, Short Form (BDI-SF)
2. Current or significant history of substance abuse
3. In the 3 months preceding enrollment, change in medications that impact neuroplasticity
4. Current participation in any other research study, cognitive rehabilitation, meditation, or mental training program, including commercial brain-training programs
5. Neurological disorder other than stroke (e.g., Parkinson's disorder; multiple sclerosis; traumatic brain injury)
6. Spatial attention deficit (unilateral neglect) defined as a score of 51 or fewer cancellations on the Star Cancellation Test.
7. According to the clinical judgement of the PI or her authorized designee, any other functional impairment which would significantly deter comprehension and/or execution of the requirements of the trial, such as aphasia, hearing deficit, or mobility deficit restricting navigation to, from, and within the research site. Subjects must be able to provide their own transportation to and from the study site.
8. Uncontrolled or severe mental or cognitive disorder with low psychosocial functioning, such as untreated schizophrenia, bipolar disorder, or autism

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-09 (Actual)

PRIMARY OUTCOMES:
Sustained Attention to Response Task, Fixed Version | through study completion; average of 4 weeks
  SARTfixed is in the class of attention tests called continuous performance tests, a class which has a long history of use to measure sustained attention (Shaleva, Ben-Simon, Mevorachc, Cohen, & Tsald, 2011). SARTfixed is a 5-minute computerized test based on the standard version of the SART, which was developed to measure sustained attention in subjects with right-hemisphere acquired brain lesions (Robertson, Manly, Andrade, Baddeley, & Yiend,1997b). Manly and colleagues (2003) demonstrated that in subjects with neurological impairment, SARTfixed was a more pure measurement of sustained attention than standard SART. SARTfixed also had comparatively more likelihood than standard SART for accurately discriminating between healthy volunteers and individuals with neurological impairment.

SECONDARY OUTCOMES:
Trail-Making Test (TMT) | through study completion; average of 4 weeks
  • TMT is a 5-minute pencil-and-paper test that has been extensively used as a measure of executive function as well as a measure of attention in a study of meditation to improve attention after stroke (Johansson, Bjuhr, & Rönnbäck, 2012).
Cognitive Failures Questionnaire | through study completion; average of 4 weeks
  • CFQ is a 25-item pencil-and-paper questionnaire that uses a self-report scale 1-5 on which subjects identify difficulty in everyday cognitive functioning. CFQ measures 4 cognitive constructs (Distractibility, Memory, Blunders and Naming) and has been used in research, as well as clinically, to measure sustained attention after stroke (Shalev, Humphreys, & Demeyere, 2016).

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Carrico, M.S., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No